CLINICAL TRIAL: NCT07315178
Title: Creation of a Digital Twin for Predicting the Progression of Patients With Chronic Thoracic Aortic Dissection
Acronym: ADEPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BOUCHOT FEDER 2024
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type A Aortic Dissection With Residual Type B Dissection; Chronic Type B Aortic Dissection
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type B aortic dissection (Experimental)
  Interventions: Other: MRI with 4D flow imaging; Biological: blood sampling
- Residual type B aortic dissection following surgery for type A aortic dissection (Experimental)
  Interventions: Other: MRI with 4D flow imaging; Biological: blood sampling

INTERVENTIONS:
Other: MRI with 4D flow imaging — At 3 months
Biological: blood sampling — 2 tubes of 10 ml blood at inclusion, at 3 months, at 12 months, at 24 months and at 36 months

SUMMARY:
Aortic dissection causes a tear in the inner layers of the aorta, leading to the formation of a true and false lumen.

There are two types of dissection: type A, which affects the ascending aorta, and type B, which affects the descending aorta. Type A aortic dissection is almost always a surgical emergency and involves replacing the ascending aorta with a prosthesis. After this type of dissection, a residual dissection remains in the descending aorta, known as residual type B dissection, which becomes chronic. This requires increased monitoring by MRI or CT scan, which are currently not effective enough to predict the development of an aneurysm that could lead to aortic rupture requiring surgical intervention. Other factors such as blood flow, the forces and mechanisms regulating blood circulation, the mechanics and histology of the aorta, and blood markers could provide a more reliable prediction of the development of an aneurysm. The creation of a digital twin model incorporating all these factors should enable better patient management.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given written consent
* Age > 18 years
* Patient with type A aortic dissection with surgical indication for replacement
* Patient with chronic type B aortic dissection, monitored and managed medically, not operated on

Exclusion Criteria:

* Persons not affiliated with or not covered by a social security scheme
* Persons subject to legal protection measures (guardianship)
* Persons subject to judicial protection measures
* Pregnant women, women in labour or breastfeeding
* Adults who are incapacitated or unable to give their consent
* Contraindications to MRI: claustrophobia, non-MRI-compatible metal implants, suspected metal foreign body
* Severe renal failure (clearance <30ml/min according to Cockroft due to gadolinium injection)
* Uncontrolled asthma
* Patients with acute type A aortic dissection who died during or in the post-operative period following surgery to repair the dissection
* Patients with a known allergy to gadolinium-based contrast agents
* Patients treated for type B aortic dissection who underwent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Relevance of combining biomarkers | 3 months, 1 year, 2 years, 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France